CLINICAL TRIAL: NCT03976375
Title: A Phase 3, Multicenter, Randomized, Open-label Trial to Compare the Efficacy and Safety of Pembrolizumab (MK-3475) in Combination With Lenvatinib (E7080/MK-7902) Versus Docetaxel in Previously Treated Participants With Metastatic Non-small Cell Lung Cancer (NSCLC) and Progressive Disease (PD) After Platinum Doublet Chemotherapy and Immunotherapy (LEAP-008)
Brief Title: Efficacy and Safety of Pembrolizumab (MK-3475) With Lenvatinib (E7080/MK-7902) vs. Docetaxel in Participants With Metastatic Non-Small Cell Lung Cancer (NSCLC) and Progressive Disease (PD) After Platinum Doublet Chemotherapy and Immunotherapy (MK-7902-008/E7080-G000-316/LEAP-008)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Collaborators: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7902-008; MK-7902-008 (Other: MSD); LEAP-008 (Other: MSD); E7080-G000-316 (Other: Eisai Inc.); 195003 (Registry Identifier: JAPIC-CTI); 2022-501439-18-00 (Registry Identifier: EU CT); U1111-1280-4337 (Registry Identifier: UTN); 2018-003791-12 (EudraCT Number)
Record Dates: First submitted 2019-06-03; First posted 2019-06-06 (Actual); Results first posted 2024-08-22 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-07

CONDITIONS: Metastatic Non-Small Cell Lung Cancer
Keywords: programmed cell death 1 (PD-1, PD1); programmed cell death-ligand 1 (PD-L1, PDL1); programmed cell death-ligand 2 (PD-L2, PDL2)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; lenvatinib; Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Pembrolizumab+Lenvatinib (Experimental): Participants receive pembrolizumab at 200 mg, every 3 weeks (Q3W) via intravenous (IV) infusion on Day 1 of each 21-day cycle, in combination with lenvatinib at 20 mg, once daily (QD) via oral capsule. Pembrolizumab will be administered for up to 35 treatment cycles (~2 years). Lenvantinib will be administered until progressive disease or unacceptable toxicity.
  Interventions: Biological: Pembrolizumab; Drug: Lenvatinib
- Docetaxel (Active Comparator): Participants receive docetaxel at 75 mg/m^2, Q3W via IV infusion over 1-hour infusion on Day 1 of each 21-day cycle. Docetaxel will be administered until progressive disease or unacceptable toxicity.
  Interventions: Drug: Docetaxel
- Lenvatinib Monotherapy (Experimental): Participants receive lenvatinib at 24 mg, QD via oral capsule. Lenvantinib will be administered until progressive disease or unacceptable toxicity.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion of pembrolizumab at 200 mg
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab+Lenvatinib
Drug: Lenvatinib — Oral capsules (unit strength: 4 and 10 mg) at 20 mg or 24 mg total daily dose.
  Other Names: MK-7902; E7080; LENVIMA®
  Arms: Lenvatinib Monotherapy; Pembrolizumab+Lenvatinib
Drug: Docetaxel — IV infusion of docetaxel at 75 mg/m^2.
  Other Names: TAXOTERE®
  Arms: Docetaxel

SUMMARY:
This study will evaluate the efficacy and safety of pembrolizumab (MK-3475) with lenvatinib (E7080/MK-7902) vs. docetaxel in participants with metastatic non-small cell lung cancer (NSCLC) and progressive disease (PD) after platinum doublet chemotherapy and treatment with one prior anti-PD-1/PD-L1 monoclonal antibody (mAb). The primary hypotheses of this study are that pembrolizumab + lenvatinib (compared with docetaxel) prolongs: 1) overall survival (OS); and progression-free survival (PFS) per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) based on blinded independent central review (BICR).

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically or cytologically confirmed diagnosis of metastatic squamous or nonsquamous Non-Small Cell Lung Cancer (NSCLC) -Stage IV: M1a, M1b, M1c.
* Has progressive disease (PD) on treatment with one prior anti-programmed cell death 1 (PD-1)/programmed cell death ligand 1 (PD-L1) monoclonal antibody (mAb) administered either as monotherapy or in combination with other checkpoint inhibitors or other therapies.

  * Retreatment with the same anti-PD-L1/PD-L1 mAb is acceptable in the overall course of treatment
* Has PD during/after platinum doublet chemotherapy for metastatic disease.
* Has confirmation that EGFR-, ALK-, or ROS1-directed therapy is not indicated as primary therapy (documentation of absence of tumor-activating EGFR mutations [eg, DEL19 or L858R], and absence of ALK and ROS1 gene rearrangements OR presence of a K-ras mutation).
* Has submitted pre-study imaging that confirmed evidence of PD following initiation of an anti-PD-1/PD-L1 inhibitor.
* Has at least 1 measurable lesion by computerized tomography (CT) or magnetic resonance imaging (MRI) per Response Evaluation Criteria in Solid Tumors (RECIST) 1.1, as determined by the local site assessment.
* Has provided tumor tissue for PD-L1 biomarker analysis from an archival sample (defined as: from initial diagnosis of NSCLC and prior to receiving immunotherapy [antiPD-1/PD-L1], from the primary lesion or a metastatic lesion).
* Has provided prior to allocation tissue from a newly obtained formalin-fixed sample from a new biopsy (defined as: after completion of immunotherapy [anti-PD-1/PD-L1] and before receiving a randomization number), of a tumor lesion not previously irradiated.
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 within 7 days before the first dose of study intervention but before randomization.
* Has a life expectancy of at least 3 months.
* Male participants receiving pembrolizumab ± lenvatinib or lenvatinib must agree to refrain from donating sperm, and either 1) be abstinent from heterosexual intercourse; or 2) follow contraceptive guidance during the treatment period or 7 days after the last dose of lenvatinib. Male participants receiving docetaxel agree to adhere to the same conditions during the treatment period and for ≥90 days after the last dose of study treatment.
* Female participants must not be pregnant, not be breastfeeding, and not be a woman of child-bearing potential (WOCBP). If a WOCBP, agrees to not donate eggs and either use contraception, or be abstinent from heterosexual intercourse during the treatment period and for ≥120 days after the last dose of pembrolizumab or 30 days after the last dose of lenvatinib, whichever occurs last. If a WOCBP receiving docetaxel, agrees to adhere to the same conditions during the treatment period and for ≥30 days after the last dose of study treatment.
* Has adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP ≤150/90 mm Hg and no change in antihypertensive medications within 1 week before randomization.
* If participant received major surgery or radiation therapy of >30 Gy, they have recovered from the toxicity and/or complications from the intervention.
* Has adequate organ function.

Exclusion Criteria:

* Has received docetaxel as monotherapy or in combination with other therapies.
* Has received lenvatinib as monotherapy or in combination with an anti-PD-1/PD-L1 mAb.
* Has received: 1) radiotherapy within 2 weeks before the first dose of study treatment; or 2) lung radiation therapy >30 Gy within 6 months before the first dose of study treatment.
* Has received a live vaccine within 30 days before the first dose of study treatment.
* Has clinically significant hemoptysis or tumor bleeding within 2 weeks before the first dose of study treatment.
* Has radiographic evidence of intratumoral cavitation, encasement, or invasion of a major blood vessel.
* Has clinically significant cardiovascular impairment within 12 months of the first dose of study treatment.
* Has a history of a gastrointestinal condition or procedure that may affect oral absorption of study treatment.
* Has a pre-existing ≥Grade 3 gastrointestinal or non-gastrointestinal fistula.
* Is currently participating in a clinical trial and receiving study therapy or participated in a study of an investigational agent within 4 weeks of the first dose of study treatment.
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days before the first dose of study treatment.
* Has a known history of an additional malignancy, except if the participant has undergone potentially curative therapy with no evidence of disease recurrence for 3 years since initiation of that therapy.
* Has known active central nervous system metastases and/or carcinomatous meningitis.
* Has severe hypersensitivity to pembrolizumab and/or any of its excipients.
* Has a sensitivity to any of the excipients contained in lenvatinib and/or docetaxel.
* Has an active autoimmune disease that has required systemic treatment in the past 2 years.
* Has a history of (noninfectious) pneumonitis that required systemic steroids or current pneumonitis/interstitial lung disease.
* Has an active infection requiring systemic therapy.
* Has a known history of human immunodeficiency virus (HIV) infection.
* Has a known history of hepatitis B reactive or known active hepatitis C virus infection.
* Has active tuberculosis.
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study.
* Is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through at least 120 days after the last dose of pembrolizumab or lenvatinib, or 90 days (male participants) or 30 days (for female participants) after the last dose of docetaxel.
* Has had an allogeneic tissue/solid organ transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 422 (Actual)
Dates: Start 2019-06-26 (Actual); Primary Completion 2023-08-11 (Actual); Study Completion 2024-08-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (143):
- United States (28):
  - Comprehensive Blood & Cancer Center [Bakersfield, CA] ( Site 1604), Bakersfield, California
  - Cancer Specialists of North Florida - Fleming Island ( Site 1675), Fleming Island, Florida
  - Mid-Florida Cancer Centers ( Site 1611), Orange City, Florida
  - University of Kentucky School of Medicine & Hospitals ( Site 1621), Lexington, Kentucky
  - Hematology Oncology Clinic ( Site 1680), Baton Rouge, Louisiana
  - Harry & Jeanette Weinberg Cancer Institute ( Site 1626), Baltimore, Maryland
  - Medstar Good Samaritan Hospital ( Site 1625), Baltimore, Maryland
  - Massachusetts General Hospital ( Site 1622), Boston, Massachusetts
  - MGH - North Shore Cancer Center ( Site 1668), Danvers, Massachusetts
  - The Mass General Cancer Center at Newton-Wellesley ( Site 1692), Newton, Massachusetts
  - University of Massachusetts Medical School ( Site 1693), Worcester, Massachusetts
  - Billings Clinic ( Site 1631), Billings, Montana
  - Bozeman Health Deaconness Cancer Center ( Site 1632), Bozeman, Montana
  - Memorial Sloan-Kettering Cancer Center At Basking Ridge ( Site 1664), Basking Ridge, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Middletown ( Site 1665), Middletown, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Montvale ( Site 1667), Montvale, New Jersey
  - Memorial Sloan-Kettering Cancer Center at Commack ( Site 1662), Commack, New York
  - Memorial Sloan-Kettering Cancer Center at West Harrison ( Site 1666), Harrison, New York
  - Memorial Sloan-Kettering Cancer Center ( Site 1661), New York, New York
  - New York Cancer and Blood Specialists ( Site 1696), Port Jefferson Station, New York
  - University of Rochester ( Site 1638), Rochester, New York
  - Memorial Sloan Kettering Cancer Center - Nassau ( Site 1670), Uniondale, New York
  - TriHealth Cancer Institute ( Site 1672), Cincinnati, Ohio
  - MetroHealth Medical Center ( Site 1694), Cleveland, Ohio
  - Kaiser Permanente Center for Health Research-Kaiser Permanente Medical Center ( Site 1644), Portland, Oregon
  - Fox Chase Cancer Center ( Site 1647), Philadelphia, Pennsylvania
  - Thompson Cancer Survival Center ( Site 1695), Knoxville, Tennessee
  - Millenium Physicians ( Site 1690), Houston, Texas
- Argentina (5):
  - Instituto de Investigaciones Metabolicas ( Site 2004), Caba, Buenos Aires
  - Hospital Britanico de Buenos Aires ( Site 2002), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Parque ( Site 2005), Rosario, Santa Fe Province
  - Hospital Aleman ( Site 2000), Buenos Aires
  - CEMIC ( Site 2003), Buenos Aires
- Australia (7):
  - Blacktown Hospital ( Site 0004), Blacktown, New South Wales
  - Port Macquarie Base Hospital ( Site 0003), Port Macquarie, New South Wales
  - Westmead Hospital ( Site 0005), Westmead, New South Wales
  - Southern Medical Day Care Centre ( Site 0001), Wollongong, New South Wales
  - Princess Alexandra Hospital - Division of Cancer Services ( Site 0002), Woolloongabba, Queensland
  - Calvary Central Districts Hospital ( Site 0007), Elizabeth Vale, South Australia
  - Bendigo Cancer Centre ( Site 0008), Bendigo, Victoria
- Canada (6):
  - CancerCare Manitoba ( Site 1504), Winnipeg, Manitoba
  - Kingston Health Sciences Centre ( Site 1503), Kingston, Ontario
  - London Regional Cancer Program - London HSC ( Site 1505), London, Ontario
  - Princess Margaret Cancer Centre ( Site 1502), Toronto, Ontario
  - CIUSSS Ouest de l Ile - St-Mary s Hospital ( Site 1501), Montreal, Quebec
  - CHUQ-Univ Laval-Hotel Dieu de Quebec ( Site 1514), Québec, Quebec
- Colombia (7):
  - Rodrigo Botero SAS ( Site 1300), Medellín, Antioquia
  - Clinica de la Costa Ltda. ( Site 1309), Barranquilla, Atlántico
  - Administradora Country SA - Clinica del Country ( Site 1307), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 1304), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 1305), Valledupar, Cesar Department
  - Oncomedica S.A. ( Site 1302), Montería, Departamento de Córdoba
  - Centro Medico Imbanaco de Cali S.A ( Site 1301), Cali, Valle del Cauca Department
- France (8):
  - CHU Caen Service de Pneumologie ( Site 0401), Caen, Calvados
  - HIA Percy-Clamart ( Site 0411), Clamart, Hauts-de-Seine
  - ICO Centre Paul Papin ( Site 0412), Angers, Maine-et-Loire
  - Clinique Ambroise Pare ( Site 0402), Beuvry, Pas-de-Calais
  - Centre Hospitalier General - Avignon ( Site 0407), Avignon, Provence-Alpes-Côte d'Azur Region
  - Centre Hospitalier Le Mans ( Site 0406), Le Mans, Sarthe
  - Institut Curie ( Site 0400), Paris
  - Hopital Europeen Georges Pompidou ( Site 0408), Paris
- Germany (4):
  - Thoraxklinik Heidelberg gGmbH am Universitaetsklinikum Heidelberg ( Site 0501), Heidelberg, Baden-Wurttemberg
  - Evangelisches Krankenhaus Hamm gGmbH ( Site 0504), Hamm, North Rhine-Westphalia
  - SRH Wald-Klinikum Gera GmbH ( Site 0503), Gera, Thuringia
  - Vivantes Klinikum Spandau ( Site 0505), Berlin
- Greece (4):
  - General Hospital of Chest Diseases "Sotiria" ( Site 1703), Athens, Attica
  - Metropolitan Hospital-4th Oncology Dept ( Site 1700), Athens, Attica
  - University Hospital of Ioannina ( Site 1701), Ioannina
  - European Interbalkan Medical Center ( Site 1704), Thessaloniki
- Hungary (9):
  - Borsod-Abaúj-Zemplén Megyei Központi Kórház és Egyetemi Oktatókórház ( Site 0601), Miskolc, Borsod-Abauj Zemplen county
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz ( Site 0606), Székesfehérvár, Fejér
  - Petz Aladar Megyei Oktato Korhaz ( Site 0609), Győr, Győr-Moson-Sopron
  - Jasz Nagykun Szolnok Megyei Hetenyi Geza Korhaz Rendelointezet ( Site 0610), Szolnok, Jász-Nagykun-Szolnok
  - Tudogyogyintezet Torokbalint ( Site 0602), Törökbálint, Pest County
  - Veszprem Megyei Tudogyogyintezet ( Site 0607), Farkasgyepű, Veszprém megye
  - Semmelweis Egyetem.. ( Site 0604), Budapest
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 0603), Budapest
  - Orszagos Koranyi Pulmonologiai Intezet ( Site 0608), Budapest
- Israel (7):
  - Soroka Medical Center ( Site 0701), Beersheba
  - Rambam Medical Center ( Site 0703), Haifa
  - Shaare Zedek Medical Center-Oncology ( Site 0706), Jerusalem
  - Meir Medical Center ( Site 0702), Kfar Saba
  - Rabin Medical Center ( Site 0700), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0704), Ramat Gan
  - Sourasky Medical Center (Ichilov) - Oncology Clinic ( Site 0705), Tel Aviv
- Italy (10):
  - Ospedale San Gerardo - ASST Monza ( Site 0804), Monza, Monza E Brianza
  - Istittuto Nazionale dei Tumori Regina Elena IRCCS - IFO ( Site 0807), Rome, Roma
  - A.O. Ospedali Riuniti Villa Sofia - Cervello P.O. Villa Sofia ( Site 0810), Palermo, Sicily
  - Ospedale San Luigi Gonzaga ( Site 0802), Orbassano, Torino
  - Azienda Ospedaliera San Giuseppe Moscati ( Site 0809), Avellino
  - IRCCS Giovanni Paolo II. Ospedale Oncologico ( Site 0808), Bari
  - AOU Policlinico Vittorio Emanuele ( Site 0811), Catania
  - Istituto Nazionale dei Tumori ( Site 0806), Milan
  - Policlinico San Matteo - Fondazione IRCCS ( Site 0812), Pavia
  - Azienda Ospedaliera di Perugia ( Site 0805), Perugia
- Japan (7):
  - Kanagawa Cardiovascular and Respiratory Center ( Site 0105), Yokohama, Kanagawa
  - Sendai Kousei Hospital ( Site 0107), Sendai, Miyagi
  - Kansai Medical University Hospital ( Site 0104), Hirakata, Osaka
  - Chiba University Hospital ( Site 0106), Chiba
  - Niigata Cancer Center Hospital ( Site 0101), Niigata
  - National Cancer Center Hospital ( Site 0103), Tokyo
  - The Cancer Institute Hospital of JFCR ( Site 0100), Tokyo
- Portugal (3):
  - Centro Hospitalar Lisboa Norte E.P.E. - Hospital Pulido Valente ( Site 1801), Lisbon
  - Hospital CUF Porto ( Site 1802), Porto
  - Inst. Portugues de Oncologia de Porto Francisco Gentil EPE ( Site 1800), Porto
- Puerto Rico (3):
  - Hematology and Oncology Institute ( Site 2105), Manatí
  - Ad-Vance Medical Research LLC ( Site 2103), Ponce
  - Puerto Rico Medical Research Center LLC ( Site 2101), San Juan
- Russia (10):
  - GBUZ Republican Clinical Oncological Dispensary ( Site 0922), Ufa, Baskortostan, Respublika
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 0918), Krasnoyarsk, Krasnoyarsk Krai
  - Main Military Clinical Hospital n.a. N.N.Burdenko ( Site 0905), Moscow, Moscow
  - Central Clinical Hospital of the Administration of the President ( Site 0910), Moscow, Moscow
  - Budgetary Healthcare Institution of Omsk Region Clinical Oncology Dispensary-Chemotherapy #1 ( Site, Omsk, Omsk Oblast
  - Railway Hospital of OJSC ( Site 0907), Saint Petersburg, Sankt-Peterburg
  - Pavlov First Saint Petersburg State Medical University ( Site 0917), Saint Petersburg, Sankt-Peterburg
  - GBUZ SPb CRPCstmc(o) ( Site 0921), Saint Petersburg, Sankt-Peterburg
  - Scientific Research Oncology Institute n.a. N.N.Petrov ( Site 0903), Saint Petersburg, Sankt-Peterburg
  - SPb SBHI City Clinical Oncological Dispensary ( Site 0901), Saint Petersburg, Sankt-Peterburg
- South Korea (4):
  - Seoul National University Bundang Hospital ( Site 0204), Seongnam-si, Kyonggi-do
  - Chungbuk National University Hospital ( Site 0201), Cheongju-si, North Chungcheong
  - Asan Medical Center ( Site 0203), Songpagu, Seoul
  - Severance Hospital Yonsei University Health System ( Site 0202), Seoul
- Spain (11):
  - Consorci Hospitalari Mataro ( Site 1008), Mataró, Barcelona
  - Hospital Universitario Marques de Valdecilla ( Site 1003), Santander, Cantabria
  - Hospital Universitario Insular de Gran Canaria ( Site 1011), Las Palmas de Gran Canaria, Las Palmas
  - Hospital Universitario Puerta de Hierro ( Site 1007), Majadahonda, Madrid
  - Hospital Universitario Quiron Madrid ( Site 1012), Pozuelo de Alarcón, Madrid
  - Hospital Central de Asturias ( Site 1002), Oviedo, Principality of Asturias
  - Hospital Clinico de Valencia ( Site 1010), Valencia, Valenciana, Comunitat
  - Hospital Universitari Vall d Hebron ( Site 1004), Barcelona
  - Hospital Ciudad de Jaen ( Site 1000), Jaén
  - Hospital Universitario Fundacion Jimenez Diaz ( Site 1005), Madrid
  - Hospital Universitario 12 de Octubre ( Site 1006), Madrid
- United Kingdom (10):
  - Hull & East Yorkshire NHS Trust. Castle Hill Hospital ( Site 1108), Cottingham, East Riding Of Yorkshire
  - Nottingham City Hospital Campus ( Site 1105), Nottingham, England
  - Leicester Royal Infirmary ( Site 1110), Leicester, Leicestershire
  - North Middlesex University Hospital NHS Trust ( Site 1109), London, London, City of
  - Guy s and St Thomas Hospital NHS Foundation Trust ( Site 1102), London, London, City of
  - Mount Vernon Cancer Centre ( Site 1107), Northwood, London, City of
  - Aberdeen Royal Infirmary ( Site 1114), Aberdeen, Scotland
  - University Hospital Coventry and Warwickshire NHS Trust ( Site 1112), Coventry, Warwickshire
  - Birmingham Heartlands Hospital ( Site 1103), Birmingham
  - St James s University Hospital ( Site 1106), Leeds

IPD SHARING:
Plan to Share IPD: Yes
https://trialstransparency.msdclinicaltrials.com/pdf/ProcedureAccessClinicalTrialData.pdf
URL: https://externaldatasharing-msd.com/

REFERENCES:
- [Result] Leighl NB, Paz-Ares L, Abreu DR, Hui R, Baka S, Bigot F, Nishio M, Smolin A, Ahmed S, Schoenfeld AJ, Daher S, Cortinovis DL, Di Noia V, Linardou H, Gainor JF, Dutcus C, Okpara CE, Deng X, Kush D, Arunachalam A, Song A, Cho BC. LEAP-008: Lenvatinib Plus Pembrolizumab for Metastatic NSCLC That Has Progressed After an Anti-Programmed Cell Death Protein 1 or Anti-Programmed Cell Death Ligand 1 Plus Platinum Chemotherapy. J Thorac Oncol. 2025 Oct;20(10):1489-1504. doi: 10.1016/j.jtho.2025.05.020. Epub 2025 Jun 3. PMID 40473109
- [Derived] Xing P, Wang M, Zhao J, Zhong W, Chi Y, Xu Z, Li J. Study protocol: A single-arm, multicenter, phase II trial of camrelizumab plus apatinib for advanced nonsquamous NSCLC previously treated with first-line immunotherapy. Thorac Cancer. 2021 Oct;12(20):2825-2828. doi: 10.1111/1759-7714.14113. Epub 2021 Aug 18. PMID 34409776
- [Derived] Taylor MH, Schmidt EV, Dutcus C, Pinheiro EM, Funahashi Y, Lubiniecki G, Rasco D. The LEAP program: lenvatinib plus pembrolizumab for the treatment of advanced solid tumors. Future Oncol. 2021 Feb;17(6):637-648. doi: 10.2217/fon-2020-0937. Epub 2020 Dec 10. PMID 33300372
- See also: Merck Clinical Trials Information — https://www.merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26246&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Groups:
- Pembrolizumab+Lenvatinib: Participants received pembrolizumab at 200 mg, every 3 weeks (Q3W) via intravenous (IV) infusion on Day 1 of each 21-day cycle, in combination with lenvatinib at 20 mg, once daily (QD) via oral capsule. Pembrolizumab is administered for up to 35 treatment cycles (~2 years). Lenvantinib is administered until progressive disease or unacceptable toxicity.
- Docetaxel: Participants received docetaxel at 75 mg/m^2, Q3W via IV infusion over 1-hour infusion on Day 1 of each 21-day cycle. Docetaxel is administered until progressive disease or unacceptable toxicity.
- Lenvatinib: Participants received lenvatinib at 24 mg, QD via oral capsule. Lenvantinib is administered until progressive disease or unacceptable toxicity.
Period: Overall Study
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel | Lenvatinib
Started | 185 | 189 | 48
Treated | 181 | 177 | 47
Completed | 0 | 0 | 0
Not Completed | 185 | 189 | 48
Not completed — Death | 158 | 160 | 42
Not completed — Lost to Follow-up | 2 | 1 | 1
Not completed — Withdrawal by Subject | 5 | 9 | 4
Not completed — Sponsor decision | 20 | 19 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel | Lenvatinib | Total
Number analyzed (Participants) | 185 | 189 | 48 | 422
Age, Continuous [Mean (Standard Deviation); unit: Years] | 64.2 (8.3) | 64.3 (9.5) | 64.0 (7.2) | 64.2 (8.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 60 | 19 | 146
  Male | 118 | 129 | 29 | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12 | 12 | 4 | 28
  Not Hispanic or Latino | 160 | 160 | 40 | 360
  Unknown or Not Reported | 13 | 17 | 4 | 34
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 2 | 0 | 5
  Asian | 22 | 32 | 8 | 62
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 3 | 0 | 5
  White | 146 | 135 | 35 | 316
  More than one race | 1 | 2 | 1 | 4
  Unknown or Not Reported | 11 | 15 | 4 | 30
Eastern Cooperative Oncology Group (ECOG) at baseline [Count of Participants; unit: Participants] — Participants were classified at baseline by ECOG Performance Status of 0 (Fully active, able to carry on all pre-disease performance without restriction) or 1 (Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature).
  Participants
    ECOG 0 | 67 | 67 | 17 | 151
    ECOG 1 | 118 | 122 | 31 | 271
Sequence of Prior Anti-programmed cell death protein 1 (PD-1)/PD-L1 Therapy [Count of Participants; unit: Participants] — Participants were classified at baseline by whether Anti-PD-1/PD-L1 was the type of therapy received immediately prior to enrollment, or not the immediate prior therapy received prior to enrollment
  Participants
    Immediate Prior Therapy -Anti-PD-1/PD-L1 | 145 | 150 | 38 | 333
    Not Immediate Prior Therapy--Anti-PD-1/PD-L1 | 40 | 39 | 10 | 89
Programmed cell death ligand 1 (PD-L1)Status [Count of Participants; unit: Participants] — Participants were stratified by PD-L1 status at baseline; Tumor proportion score (TPS) <50% or TPS>=50%
  Participants
    TPS<50% | 135 | 140 | 34 | 309
    TPS>=50% | 34 | 33 | 10 | 77
    Unknown | 16 | 16 | 4 | 36

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS is defined as the time from randomization to the date of death due to any cause.
Time Frame: Up to ~47 months
Population: All randomized participants, included in the treatment group to which they were randomized. Per protocol, participants in the lenvatinib monotherapy arm were not analyzed.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Lenvatinib Monotherapy: Participants received lenvatinib at 24 mg, QD via oral capsule. Lenvatinib is administered until progressive disease or unacceptable toxicity.
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel | Lenvatinib Monotherapy
Number analyzed (Participants) | 185 | 189 | 0
Months | 11.3 [9.4 to 13.2] | 12.0 [9.6 to 13.7] |
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Superiority; p = 0.4342, Log Rank — Stratified by Baseline ECOG performance status (0 versus 1), anti-PD-1/PD-L1 mAb (immediate prior therapy versus not the immediate prior therapy), and Baseline PD-L1 Status (<50% versus >=50); Hazard Ratio (HR) = 0.98, 95% CI 2-sided [0.78 to 1.23] — Based on stratified Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by Baseline ECOG performance status, anti-PD-1/PD-L1 mAb therapy, and Baseline PD-L1 Status

2. Primary Outcome: Progression-free Survival (PFS) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: PFS is defined as the time from randomization to the first documented progressive disease (PD) or death due to any cause, whichever occurs first. Per RECIST 1.1, PD is defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of ≥5 mm. Note: The appearance of one or more new lesions is also considered PD. PFS was assessed by blinded independent central review (BICR) per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Time Frame: Up to ~47 months
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel | Lenvatinib Monotherapy
Number analyzed (Participants) | 185 | 189 | 0
Months | 5.6 [4.2 to 6.5] | 4.2 [3.2 to 5.2] |
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Superiority; p = 0.1563, Log Rank — [p-value comment as in outcome 1, analysis 1]; Hazard Ratio (HR) = 0.89, 95% CI 2-sided [0.70 to 1.12] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) - Pembrolizumab+Lenvatinib vs. Docetaxel
Description: ORR is defined as the percentage of participants who have a Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions). ORR was assessed by BICR per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Time Frame: Up to ~47 months
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel | Lenvatinib Monotherapy
Number analyzed (Participants) | 185 | 189 | 0
Percentage of Participants | 22.7 [16.9 to 29.4] | 14.3 [9.6 to 20.1] |
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Superiority; p = 0.01818, Miettinen and Nurminen method — One-sided p-value for testing. H0: difference in % =0 versus H1: difference in % > 0; Difference in Percentage vs Docetaxel = 8.4, 95% CI 2-sided [0.5 to 16.3] — Based on Miettinen & Nurminen method stratified by Baseline ECOG performance status (0 versus 1), anti-PD-1/PD-L1 mAb (immediate prior therapy versus not the immediate prior therapy), and Baseline PD-L1 Status (<50% versus >=50%)

4. Secondary Outcome: Objective Response Rate (ORR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) - Pembrolizumab+Lenvatinib vs. Lenvatinib Monotherapy
Description: as for outcome 3
Time Frame: Up to ~47 months
Population: All randomized participants, included in the treatment group to which they were randomized. Per protocol, participants in the docetaxel arm were not analyzed.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab+Lenvatinib | Lenvatinib Monotherapy | Docetaxel
Number analyzed (Participants) | 185 | 48 | 0
Percentage of Participants | 22.7 [16.9 to 29.4] | 12.5 [4.7 to 25.2] |
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Lenvatinib Monotherapy; Test type: Superiority; p = 0.06009, Miettinen & Nurminen method — One-sided p-value for testing. H0: difference in % =0 versus H1: difference in % > 0; Difference in Percentage vs Lenvatinib = 10.2, 95% CI 2-sided [-3.1 to 19.9]

5. Secondary Outcome: Duration of Response (DOR) Per Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1)
Description: DOR is defined as the time from first documented evidence of Complete Response (CR: Disappearance of all target lesions) or a Partial Response (PR: At least a 30% decrease in the sum of diameters of target lesions) until disease progression or death due to any cause, whichever occurs first. DOR was assessed by BICR per RECIST 1.1, modified to follow a maximum of 10 target lesions and a maximum of 5 target lesions per organ.
Time Frame: Up to ~47 months
Population: All randomized participants who had a confirmed or partial response, included in the treatment group to which they were randomized. Per protocol, participants in the lenvatinib monotherapy arm were not analyzed.
Measure: Median (Full Range); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel | Lenvatinib Monotherapy
Number analyzed (Participants) | 42 | 27 | 0
Months | 6.9 [2.3 to NA] — NA= Upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse | 6.8 [NA to NA] — NA= lower limit, upper limit not reached at time of data cut-off due to insufficient number of responding participants with relapse |

6. Secondary Outcome: Number of Participants Experiencing an Adverse Event (AE)
Description: An AE is any untoward medical occurrence in a clinical study participant that is temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experienced an AE is presented.
Time Frame: Up to ~47 months
Population: All randomized participants who received at least 1 dose of study intervention
Measure: Number; unit: Participants
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel | Lenvatinib Monotherapy
Number analyzed (Participants) | 181 | 177 | 47
Participants | 179 | 174 | 47

7. Secondary Outcome: Number of Participants Discontinuing Study Treatment Due to an AE
Description: The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to ~47 months
Population: All randomized participants who received at least 1 dose of study intervention
Measure: Number; unit: Participants
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel | Lenvatinib Monotherapy
Number analyzed (Participants) | 181 | 177 | 47
Participants | 68 | 43 | 13

8. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment (EORTC) Quality of Life Questionnaire-Core 30 (QLQ-C30) Combined Global Health Status / Quality of Life (Items 29 & 30) Scale Combined Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the quality of life (QoL) of cancer patients, including a combined global health status (GHS)/QoL (Items 29 and 30) scale. For each item, scores range from 0-100, with higher scores indicating higher GHS/QoL. Per protocol, scores for items 29 and 30 will be averaged to compute a combined GHS/QoL scale score. Change from baseline in the combined GHS/QoL scale scores is presented.
Time Frame: Baseline and Week 12
Population: Randomized participants in pembrolizumab + lenvatinib and docetaxel arms, who have at least 1 EORTC QLQ-C30 assessment available and have received at least 1 dose of study intervention. Participants were analyzed in the treatment group to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel
Number analyzed (Participants) | 181 | 176
Scores on a scale | -2.48 [-5.44 to 0.49] | -1.12 [-4.22 to 1.98]
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Other; p = 0.4998, t-test, 2 sided; Difference in least squares means = -1.36, 95% CI 2-sided [-5.32 to 2.60] — Based on cLDA model with covariates for treatment by time interaction, stratification factors of baseline ECOG performance status, anti-PD-1/PD-L1 mAb therapy, and baseline PD-L1 Status

9. Secondary Outcome: Change From Baseline in EORTC Quality of Life Questionnaire Lung Cancer Module 13 (QLQ-LC13) Cough (Item 31) Scale Score
Description: Used in combination with QLQ-C30, the EORTC QLQ-LC13 is a supplemental lung cancer-specific module, including a single-item scale score for cough (Item 31). For this item, individual responses to the question "How much did you cough?" are given on a 4-point scale (1=Not at all; 4=Very much). Scores are transformed to a range from 0-100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-LC13 cough (Item 31) scale score is presented.
Time Frame: Baseline and Week 12
Population: Randomized participants in pembrolizumab + lenvatinib and docetaxel arms, who have at least 1 EORTC QLQ-LC13 assessment available and have received at least 1 dose of study intervention. Participants were analyzed in the treatment group to which they were randomized.
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel
Number analyzed (Participants) | 181 | 175
Scores on a scale | -4.17 [-8.08 to -0.27] | -0.32 [-4.40 to 3.77]
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Other; p = 0.1531, t-test, 2 sided; Difference in Least Squares Mean = -3.86, 95% CI 2-sided [-9.16 to 1.44] — [estimate comment as in outcome 8, analysis 1]

10. Secondary Outcome: Change From Baseline in EORTC QLQ-LC13 Chest Pain (Item 40) Scale Score
Description: Used in combination with QLQ-C30, the EORTC QLQ-LC13 is a supplemental lung cancer-specific module, including a single-item scale score for chest pain (Item 40). For this item, individual responses to the question "Have you had pain in your chest?" are given on a 4-point scale (1=Not at all; 4=Very much). Scores are transformed to a range from 0-100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-LC13 chest pain (Item 40) scale score is presented.
Time Frame: Baseline and Week 12
Population: as for outcome 9
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel
Number analyzed (Participants) | 181 | 175
Scores on a scale | -1.40 [-4.92 to 2.12] | -3.88 [-7.58 to -0.18]
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Other; p = 0.3084, t-test, 2 sided; Difference in Least Squares Means = 2.48, 95% CI 2-sided [-2.31 to 7.27] — Based on cLDA model with covariates for treatment by time interaction, stratification factors of baseline ECOG performance status, timing of anti-PD-1/PD-L1 mAb therapy, and baseline PD-L1 Status

11. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Dyspnea (Item 8) Scale Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients, including a single-item scale score for dyspnea (Item 8). For this item, individual responses to the question "Were you short of breath?" are given on a 4-point scale (1=Not at all; 4=Very much). Scores are transformed to a range from 0-100, with a lower score indicating a better outcome. The change from baseline in the EORTC QLQ-C30 dyspnea (Item 8) scale score is presented.
Time Frame: Baseline and Week 12
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel
Number analyzed (Participants) | 181 | 176
Scores on a scale | -2.92 [-7.08 to 1.23] | 5.12 [0.79 to 9.45]
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Other; p = 0.0058, t-test, 2 sided; Difference in Least Squares Means = -8.04, 95% CI 2-sided [-13.73 to -2.35] — [estimate comment as in outcome 8, analysis 1]

12. Secondary Outcome: Change From Baseline in EORTC QLQ-C30 Physical Functioning (Items 1 to 5) Scale Combined Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients, including a physical functioning (PF) scale (Items 1 to 5). The PF scale consists of participant responses to 5 questions regarding performance of daily activities [1) strenuous activities; 2) long walks; 3) short walks; 4) bed/chair rest; and 5) needing help with eating, dressing, washing themselves or using the toilet]. Overall PF scores range from 0 to 100, with a lower score indicating a better outcome. The change from Baseline in the EORTC QLQ-C30 PF (Items 1 to 5) scale combined score is presented.
Time Frame: Baseline and Week 12
Population: as for outcome 8
Measure: Least Squares Mean (95% Confidence Interval); unit: Scores on a scale
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel
Number analyzed (Participants) | 181 | 176
Scores on a scale | -5.58 [-8.51 to -2.65] | -8.47 [-11.51 to -5.43]
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Other; p = 0.1681, t-test, 2 sided; Difference in Least Squares Means = 2.89, 95% CI 2-sided [-1.23 to 7.01] — [estimate comment as in outcome 8, analysis 1]

13. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-C30 Combined Global Health Status / Quality of Life (Items 29 & 30) Scale Combined Score
Description: The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients, including a combined GHS/QoL (Items 29 and 30) scale. The TTD in the combined GHS/QoL (Items 29 & 30) scale combined score is presented, defined as the time to first onset of a ≥10 point decrease from baseline. A longer TTD indicates a better outcome
Time Frame: Up to 24 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel
Number analyzed (Participants) | 175 | 167
Months | 8.51 [6.24 to NA] — NA= Upper limit not reached | 9.59 [5.78 to NA] — NA=Upper limit not reached
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Other; p = 0.6145, Log Rank — stratified by Baseline ECOG performance status, anti-PD-1/PD-L1 mAb therapy, and Baseline PD-L1 Status; Hazard Ratio (HR) = 0.91, 95% CI 2-sided [0.63 to 1.31] — [estimate comment as in outcome 1, analysis 1]

14. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-LC13 Cough (Item 31) Scale Score
Description: Used in combination with QLQ-C30, the EORTC QLQ-LC13 is a supplemental lung cancer-specific module, including a single-item scale score for cough (Item 31). The TTD in EORTC QLQ-LC13 cough (Item 31) scale score is presented, defined as the time to first onset of a ≥10 point decrease from baseline.
Time Frame: Up to ~24 months
Population: as for outcome 9
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel
Number analyzed (Participants) | 173 | 164
Months | NA [NA to NA] — NA=median, lower limit and upper limit not reached | NA [10.97 to NA] — NA=median, upper limit not reached
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Other; p = 0.0398, Log Rank; Stratified by Baseline ECOG performance status, anti-PD-1/PD-L1 mAb therapy, and Baseline PD-L1 Status; Hazard Ratio (HR) = 0.61, 95% CI 2-sided [0.38 to 0.98] — [estimate comment as in outcome 1, analysis 1]

15. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-LC13 Chest Pain (Item 40) Scale Score
Description: Used in combination with QLQ-C30, the EORTC QLQ-LC13 is a supplemental lung cancer-specific module, including a single-item scale score for chest pain (Item 40). The TTD in EORTC QLQ-LC13 chest pain (Item 40) scale score is presented, defined as the time to first onset of a ≥10 point decrease from baseline.
Time Frame: Up to ~24 months
Population: Randomized participants in pembrolizumab + lenvatinib and docetaxel arms. who have at least 1 EORTC QLQ-LC13 assessment available and have received at least 1 dose of study intervention. Participants were analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel
Number analyzed (Participants) | 173 | 164
Months | NA [NA to NA] — NA= median, lower limit, upper limit not reached | NA [NA to NA] — NA= median, lower limit, upper limit not reached
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Other; p = 0.8724, Log Rank; Stratified by Baseline ECOG performance status, anti-PD-1/PD-L1 mAb therapy, and Baseline PD-L1 Status; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.59 to 1.85] — [estimate comment as in outcome 1, analysis 1]

16. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-C30 Dyspnea (Item 8) Scale Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients, including a single-item scale score for dyspnea (Item 8). The TTD in dyspnea (Item 8) scale score will be presented, defined as the time to first onset of a ≥10 point decrease from baseline.
Time Frame: Up to ~24 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel
Number analyzed (Participants) | 175 | 167
Months | NA [NA to NA] — NA=median, lower limit, upper limit not reached | NA [10.84 to NA] — NA=Median, upper limit not reached
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Other; p = 0.1944, Log Rank — Stratified by Baseline ECOG performance status, anti-PD-1/PD-L1 mAb therapy, and Baseline PD-L1 Status; Hazard Ratio (HR) = 0.75, 95% CI 2-sided [0.49 to 1.16] — [estimate comment as in outcome 1, analysis 1]

17. Secondary Outcome: Time to True Deterioration (TTD) in EORTC QLQ-C30 Physical Functioning (Items 1 to 5) Scale Combined Score
Description: The EORTC QLQ-C30 is a 30-item questionnaire developed to assess the QoL of cancer patients, including a physical functioning (PF) scale (Items 1 to 5). The TTD in PF (Items 1 to 5) scale combined score is presented, defined as the time to first onset of a ≥10 point decrease from baseline.
Time Frame: Up to ~24 months
Population: as for outcome 8
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel
Number analyzed (Participants) | 175 | 167
Months | 6.70 [5.36 to 9.86] | 7.03 [4.76 to NA] — NA=upper limit not reached
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Other; p = 0.9837, Log Rank; Stratified by Baseline ECOG performance status, anti-PD-1/PD-L1 mAb therapy, and Baseline PD-L1 Status; Hazard Ratio (HR) = 1.00, 95% CI 2-sided [0.71 to 1.41] — [estimate comment as in outcome 1, analysis 1]

18. Secondary Outcome: Time to True Deterioration (TTD) in EORTC Composite Symptom Score for Cough (QLQ-LC13 Item 31), Chest Pain (QLQ-LC13 Item 40), or Dyspnea (QLQ-C30 Item 8)
Description: EORTC QLQ-C30 includes a single-item scale score for dyspnea (Item 8), the EORTC QLQ-LC13 is a supplemental lung cancer-specific module, which includes a single-item scale score for cough (Item 31) and chest pain (Item 40). Time to True Deterioration for the Composite Endpoint of EORTC QLQ- LC13 Cough, EORTC QLQ- LC13 Chest Pain, or EORTC QLQ-C30 Dyspnea is presented, defined as the time to first onset of a ≥10-point decrease from baseline in any one of 3 scale items with confirmation by the subsequent visit of a 10 or more-point deterioration from baseline in the same scale as the first onset under right-censoring rule.
Time Frame: Up to ~ 24 months
Population: Randomized participants in pembrolizumab + lenvatinib and docetaxel arms, who have at least 1 EORTC QLQ-C30 and EORTC QLC-LC13 assessment available and have received at least 1 dose of study intervention. Participants were analyzed in the treatment group to which they were randomized.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab+Lenvatinib | Docetaxel
Number analyzed (Participants) | 175 | 167
Months | 9.20 [5.59 to 12.62] | 5.55 [3.48 to 12.78]
Statistical Analysis 1: Comparison: Pembrolizumab+Lenvatinib vs Docetaxel; Test type: Other; p = 0.2903, Log Rank; Stratified by Baseline ECOG performance status, anti-PD-1/PD-L1 mAb therapy, and Baseline PD-L1 Status; Hazard Ratio (HR) = 0.84, 95% CI 2-sided [0.60 to 1.16] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Up to approximately 59 months
Description: The population for all-cause mortality includes all participants in the treatment arm to which they were randomized. SAE and other AEs population includes all randomized participants who received at least 1 dose of study intervention. MedDRA preferred terms 'Neoplasm progression' 'Malignant neoplasm progression' and 'Disease progression' not related to the drug are excluded.
Groups:
- Pembrolizumab + Lenvatinib: Participants received pembrolizumab at 200 mg, every 3 weeks (Q3W) via intravenous (IV) infusion on Day 1 of each 21-day cycle, in combination with lenvatinib at 20 mg, once daily (QD) via oral capsule. Pembrolizumab is administered for up to 35 treatment cycles (~2 years). Lenvantinib is administered until progressive disease or unacceptable toxicity.
- Lenvatinib: Participants received lenvatinib at 24 mg, QD via oral capsule. Lenvatinib is administered until progressive disease or unacceptable toxicity.
Arm/Group | Pembrolizumab + Lenvatinib | Docetaxel | Lenvatinib
All-Cause Mortality (participants affected / at risk) | 161/185 | 164/189 | 46/48
Serious Adverse Events (participants affected / at risk) | 99/181 | 66/177 | 28/47
Other Adverse Events (participants affected / at risk) | 170/181 | 165/177 | 45/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenvatinib (N=181) | Docetaxel (N=177) | Lenvatinib (N=47)
Agranulocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 1 (2) | 1 (1)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 8 (8) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Angina pectoris (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Angina unstable (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (2) | 0 (0) | 0 (0)
Atrioventricular block complete (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 2 (2) | 2 (2) | 3 (3)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 3 (3) | 2 (2) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 2 (2) | 0 (0) | 0 (0)
Left ventricular dysfunction (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2) | 1 (1) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 1 (1) | 1 (1)
Hypoaldosteronism (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Hypophysitis (Endocrine disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Anal inflammation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 4 (4) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 7 (7) | 2 (2) | 0 (0)
Duodenal ulcer (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastric perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0)
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Haematemesis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Large intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Small intestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Asthenia (General disorders) | 2 (2) | 2 (2) | 1 (1)
Condition aggravated (General disorders) | 0 (0) | 0 (0) | 1 (1)
Death (General disorders) | 2 (2) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 1 (1) | 0 (0) | 0 (0)
General physical health deterioration (General disorders) | 1 (1) | 1 (1) | 0 (0)
Inadequate analgesia (General disorders) | 0 (0) | 1 (1) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 3 (4) | 2 (2) | 0 (0)
Sudden death (General disorders) | 1 (1) | 0 (0) | 0 (0)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholangitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder enlargement (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1)
Jaundice (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Abdominal sepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Anal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Biliary sepsis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Bronchopulmonary aspergillosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 2 (2) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Cholecystitis infective (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Empyema (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Escherichia infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 3 (3)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 4 (4) | 0 (0)
Oral candidiasis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Orchitis (Infections and infestations) | 0 (0) | 1 (2) | 0 (0)
Paronychia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 10 (12) | 9 (10) | 2 (2)
Postoperative wound infection (Infections and infestations) | 1 (3) | 0 (0) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 2 (2) | 0 (0)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Scrotal abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 2 (2) | 1 (1)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 2 (2) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Delayed effects of radiation (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Extradural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (3) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Radiation necrosis (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Tracheal haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Wound dehiscence (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
General physical condition abnormal (Investigations) | 0 (0) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 1 (1) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 4 (7) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 1 (1)
Autoimmune encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Encephalitis toxic (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Haemorrhage intracranial (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Neuralgia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
Posterior reversible encephalopathy syndrome (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Toxic leukoencephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Urinary tract obstruction (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1) | 0 (0)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0) | 0 (0)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 0 (0)
Hydrothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Malignant pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) | 0 (0)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 2 (2) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (2) | 2 (2)
Pulmonary haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1)
Hidradenitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Subcutaneous emphysema (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Dry gangrene (Vascular disorders) | 0 (0) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 4 (4) | 0 (0) | 0 (0)
Hypertensive crisis (Vascular disorders) | 0 (0) | 0 (0) | 2 (2)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Lenvatinib (N=181) | Docetaxel (N=177) | Lenvatinib (N=47)
Anaemia (Blood and lymphatic system disorders) | 23 (25) | 50 (56) | 2 (2)
Neutropenia (Blood and lymphatic system disorders) | 1 (5) | 9 (10) | 0 (0)
Hyperthyroidism (Endocrine disorders) | 8 (9) | 1 (1) | 3 (3)
Hypothyroidism (Endocrine disorders) | 64 (74) | 3 (3) | 17 (17)
Abdominal pain (Gastrointestinal disorders) | 26 (34) | 5 (5) | 9 (10)
Abdominal pain upper (Gastrointestinal disorders) | 15 (18) | 3 (3) | 4 (6)
Constipation (Gastrointestinal disorders) | 27 (33) | 16 (19) | 12 (13)
Diarrhoea (Gastrointestinal disorders) | 74 (133) | 35 (44) | 18 (38)
Dry mouth (Gastrointestinal disorders) | 5 (5) | 2 (2) | 7 (7)
Dyspepsia (Gastrointestinal disorders) | 15 (16) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 40 (56) | 33 (37) | 16 (21)
Stomatitis (Gastrointestinal disorders) | 32 (39) | 19 (21) | 10 (13)
Vomiting (Gastrointestinal disorders) | 31 (45) | 19 (23) | 12 (20)
Asthenia (General disorders) | 50 (61) | 47 (54) | 12 (14)
Chest pain (General disorders) | 12 (12) | 6 (7) | 6 (6)
Fatigue (General disorders) | 42 (54) | 38 (47) | 16 (18)
Oedema peripheral (General disorders) | 17 (19) | 26 (26) | 3 (4)
Pyrexia (General disorders) | 10 (11) | 33 (46) | 2 (2)
Urinary tract infection (Infections and infestations) | 15 (17) | 6 (6) | 7 (10)
Fall (Injury, poisoning and procedural complications) | 3 (4) | 1 (1) | 4 (4)
Alanine aminotransferase increased (Investigations) | 19 (26) | 7 (11) | 2 (4)
Amylase increased (Investigations) | 17 (20) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 19 (33) | 6 (10) | 2 (4)
Blood alkaline phosphatase increased (Investigations) | 15 (18) | 4 (5) | 2 (2)
Blood creatinine increased (Investigations) | 17 (21) | 3 (6) | 1 (1)
Blood thyroid stimulating hormone increased (Investigations) | 23 (28) | 0 (0) | 3 (5)
Lipase increased (Investigations) | 14 (17) | 5 (6) | 3 (4)
Neutrophil count decreased (Investigations) | 9 (11) | 36 (63) | 3 (3)
Platelet count decreased (Investigations) | 26 (30) | 4 (4) | 6 (6)
Weight decreased (Investigations) | 35 (37) | 9 (9) | 10 (10)
White blood cell count decreased (Investigations) | 2 (5) | 14 (20) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 57 (68) | 36 (38) | 13 (16)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 10 (11) | 8 (9) | 3 (3)
Hypokalaemia (Metabolism and nutrition disorders) | 17 (25) | 9 (10) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 14 (17) | 7 (8) | 3 (3)
Hyponatraemia (Metabolism and nutrition disorders) | 11 (16) | 7 (13) | 3 (5)
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 (36) | 11 (13) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 16 (17) | 10 (10) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 (4) | 2 (2) | 4 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 16 (16) | 20 (23) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (14) | 10 (11) | 4 (4)
Dizziness (Nervous system disorders) | 19 (22) | 11 (12) | 5 (6)
Dysgeusia (Nervous system disorders) | 11 (11) | 7 (9) | 3 (3)
Headache (Nervous system disorders) | 20 (27) | 5 (6) | 6 (10)
Lethargy (Nervous system disorders) | 3 (3) | 2 (2) | 3 (3)
Neuropathy peripheral (Nervous system disorders) | 4 (4) | 15 (19) | 0 (0)
Paraesthesia (Nervous system disorders) | 2 (2) | 14 (14) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 12 (15) | 1 (1)
Proteinuria (Renal and urinary disorders) | 36 (50) | 0 (0) | 7 (14)
Cough (Respiratory, thoracic and mediastinal disorders) | 27 (28) | 14 (16) | 5 (6)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 21 (26) | 5 (7) | 9 (11)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 24 (25) | 24 (24) | 7 (8)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 14 (16) | 2 (2) | 3 (5)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 14 (24) | 8 (9) | 3 (5)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (10) | 4 (5) | 3 (6)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 3 (3)
Alopecia (Skin and subcutaneous tissue disorders) | 3 (3) | 46 (46) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 8 (8) | 5 (5) | 6 (6)
Nail discolouration (Skin and subcutaneous tissue disorders) | 1 (1) | 10 (10) | 0 (0)
Nail disorder (Skin and subcutaneous tissue disorders) | 0 (0) | 9 (9) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 12 (14) | 4 (4) | 4 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 23 (30) | 9 (9) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 20 (31) | 7 (7) | 4 (4)
Hypertension (Vascular disorders) | 75 (128) | 6 (7) | 24 (34)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-12-08): https://cdn.clinicaltrials.gov/large-docs/75/NCT03976375/Prot_SAP_001.pdf